CLINICAL TRIAL: NCT01989273
Title: Detection and Management of Non-Compressible Hemorrhage by Vena Cava Ultrasonography
Status: Completed | Type: Observational
Sponsor: University of California, San Diego (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency); Emory University (Other); University of Utah (Other); Virginia Commonwealth University (Other)
Responsible Party: Principal Investigator, Jay Doucet, Professor of Surgery, University of California, San Diego
Other Study IDs: NTI-NCH-10-016; NTI W81XWH-15-1-0709 (Other Grant/Funding Number: National Trauma Institute)
Record Dates: First submitted 2013-11-14; First posted 2013-11-20 (Estimated); Last update posted 2018-07-11 (Actual); Status verified 2018-07

CONDITIONS: Trauma; Wounds and Injuries
Keywords: Trauma; Ultrasound; Shock; Resuscitation
MeSH Terms: conditions — Wounds and Injuries; Shock

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- IVC Collapsibility >50% or IVC < 12mm: Major Trauma Victims admitted at Level I Trauma Center with an inferior vena cava collapsibility >50% or IVC diameter less than or equal to 12mm
  Interventions: Device: Ultrasound of inferior vena cava
- IVC Collapsibility <50% or IVC >12mm: Major Trauma Victims admitted at Level I Trauma Center with an inferior vena cava collapsibility <50% or IVC diameter >12mm
  Interventions: Device: Ultrasound of inferior vena cava

INTERVENTIONS:
Device: Ultrasound of inferior vena cava

SUMMARY:
This is a study of patients admitted with major traumatic injuries. Such patients may develop inadequate circulation to the organs as a result of internal blood loss. Early detection of internal blood loss can be difficult as physical examination alone may miss patients with significant blood loss. Some patients with internal bleeding will arrive with low blood pressure; these patients are usually given 2 liters of intravenous fluid to determine if their blood pressure will recover. If the blood pressure does not rise or if it drops again later, the blood loss can be assumed to be severe, and the patient will likely need transfusions, surgery and other interventions. However, this fluid treatment method can lead to delays and complications as some patients may initially respond but then continue to bleed. The inferior vena cava (IVC) is the large vein draining blood from the lower body to the heart. The inferior vena cava is known to empty when the patient has had significant blood loss. The vena cava diameter can be seen using ultrasound. This study intends to perform ultrasound to examine the vena cava diameter on patients just after arriving with major trauma. The hypothesis of the proposed study is that an ultrasound assessment protocol of inferior vena cava diameter and collapsibility can detect and aid management of non-compressible hemorrhage in major trauma victims. After the patient has been given the 2 liter intravenous fluid treatment, the inferior vena cava diameter will be measured again. A third examination 8-24 hours after admission will determine if the inferior vena cava diameter has returned to normal. We propose that measuring the inferior vena cava in this manner can predict those patients who are likely to continue bleeding and require interventions such as surgery. Early detection in these patients may avoid delays in treatment, complications and excess mortality. Because this examination is done with handheld ultrasound machines, it could be done outside hospitals and in military combat casualty care.

ELIGIBILITY:
Inclusion Criteria:

* Major trauma patients brought to Level I Trauma Centers.
* Selected patients for the study will be those presenting with IVC collapsibility > 50% on modified-FAST at admission and/or
* IVC diameter of < 12mm on modified FAST at admission and/or
* A non-visualized IVC due to total collapse on modified FAST at admission (not due to body habitus or inadequate ultrasonography technique)

Exclusion Criteria:

* Pregnancy after 20 weeks gestation
* Those under 18 years of age
* Prisoners and others prohibited from participating in clinical trials
* Patients with severe traumatic brain injury who at admission are deemed by treating surgeons as having non-survivable brain injuries

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted as Major Trauma Victims via Emergency Medical Services to Level 1 Trauma Centers
Sampling Method: Non-Probability Sample
Enrollment: 121 (Actual)
Dates: Start 2012-08; Primary Completion 2018-03-01 (Actual); Study Completion 2018-03-01 (Actual)

PRIMARY OUTCOMES:
All Cause Mortality | 30 Day

SECONDARY OUTCOMES:
Need for hemostatic intervention | 30 day
Need for blood product transfusions | 30 day

CONTACTS AND LOCATIONS:
Overall Officials: Jay J Doucet, MD, Principal Investigator — University of California, San Diego
Locations (5):
- United States (5):
  - University of California San Diego Health System, San Diego, California
  - Emory University, Atlanta, Georgia
  - University of Maryland, Shock Trauma, Baltimore, Maryland
  - University of Utah, Salt Lake City, Utah
  - Virginia Commonwealth University, Richmond, Virginia

REFERENCES:
- [Derived] Doucet JJ, Ferrada P, Murthi S, Nirula R, Edwards S, Cantrell E, Han J, Haase D, Singleton A, Birkas Y, Casola G, Coimbra R; AAST Multi-Institutional Trials Committee. Ultrasonographic inferior vena cava diameter response to trauma resuscitation after 1 hour predicts 24-hour fluid requirement. J Trauma Acute Care Surg. 2020 Jan;88(1):70-79. doi: 10.1097/TA.0000000000002525. PMID 31688824